CLINICAL TRIAL: NCT04848792
Title: Treatment Strategy to Enhance Nrf2 Signaling in Older Adults: Combining Acute Exercise With the Phytochemical Sulforaphane
Brief Title: Treatment Strategy to Enhance Nrf2 Signaling in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Arizona University (Other)
Collaborators: Villanova University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1551363
Record Dates: First submitted 2021-03-16; First posted 2021-04-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Aging Problems
Keywords: Redox; Sulforaphane; Nrf2; Exercise
MeSH Terms: conditions — Motor Activity | interventions — sulforaphane

STUDY DESIGN:
Intervention Model Description: Humans
Who Masked: Participant, Investigator
Masking Description: The design of this experiment will be a randomized, double-blind, placebo-controlled, cross-over design, where each subject will serve as their own control. Randomization of order of trials (supplement/placebo) will be performed by a person that is otherwise not part of study personnel, and study personnel and subjects will be blinded to the order. The person doing the randomizing will keep a record of the order using study ID, and researchers will be unblinded upon completion of data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFN supplement (Experimental): The oral sulforaphane supplement is a myrosinase-active whole broccoli sprout material (EnduraCell Bioactive, Cell-Logic, Queensland, AU) containing 14 mg SFN per capsule. Three capsules will be consumed 90 min prior to the start of the acute exercise trial. The dose of 3 capsules is equivalent to approximately 220 µmol of SFN, which is comparable to that of other studies using broccoli sprout extracts and the recommended single dose.
  Interventions: Dietary Supplement: Sulforaphane; Dietary Supplement: Placebo capsules
- Placebo (Placebo Comparator): Placebo capsules provided by Cell-Logic.
  Interventions: Dietary Supplement: Sulforaphane; Dietary Supplement: Placebo capsules

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Myrosinase-active whole broccoli sprout material
  Other Names: EnduraCell Bioactive
Dietary Supplement: Placebo capsules — Placebo capsules

SUMMARY:
Exercise is the cornerstone of disease prevention and often an important component of treatment. However, the efficacy of an exercise stimulus is reduced with aging. This study will investigate whether adding a treatment with phytonutrients found in cruciferous vegetables can improve the exercise response in older individuals.

DETAILED DESCRIPTION:
Redox balance plays a key role in the age-associated increased risk for diseases. One reason for the lower resistance to oxidative stress with age is a gradual shift in the redox state toward a more oxidized cellular environment resulting in disruption of cell signaling. Nuclear erythroid factor 2-related factor 2 (Nrf2) is the master regulator of antioxidant defenses. Nrf2 drives expression of a host of genes involved in cytoprotection and antioxidant defenses. The Traustadottir lab was the first to demonstrate Nrf2 activation in response to acute exercise in humans, and in agreement with animal data, found an age-related impairment in exercise-induced Nrf2 signaling. This underscores an important problem related to aging, namely that older individuals are less sensitive to an exercise stimulus compared to younger cohorts. The focus of the proposed study is to try to solve this problem by amplifying the signal and mitigating the "exercise desensitization" exhibited by older individuals to restore redox balance. This study will test the hypothesis that combining acute exercise with sulforaphane will improve Nrf2 activation and downstream signaling in older adults compared to either alone. Sulforaphane (SFN) is a phytonutrient found in high concentrations in cruciferous vegetables and a potent Nrf2 activator. The hypothesis will be tested using two different approaches; the first experiment will use an in vivo-ex vivo approach, where peripheral blood mononuclear cells (PBMCs) collected from older men and women (≥60y, n=30) pre- and post-acute exercise (in vivo) will be cultured and stimulated with SFN (ex vivo). This allows for a greater experimental control of the SFN stimulus. The second experiment will test the clinical translation applying the sulforaphane stimulus in vivo through an oral supplementation of sulforaphane in the form of whole broccoli sprout material, prior to acute exercise, in the same individuals. This second experiment will be a randomized placebo-controlled cross-over design. For all trials Nrf2 signaling will be measured by Nrf2 activation through an ARE binding assay, nuclear to whole cell ratio of Nrf2 protein, and Nrf2-dependent gene expression (HO-1, GCLC, NQO1, GR). Potential sex differences will be investigated. The insights gained from this study are whether combining simple interventions in the category of healthy lifestyle and preventive medicine can improve the adaptive response to exercise in older individuals. This could have an enormous impact by improving the health and well-being of older Americans.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 60 years and older
* Competent to independently give informed consent
* Successful completion of screening
* Maximal oxygen consumption below the 60th percentile based on gender:
* Women: ≤ 21.2 mL/kg/min
* Men: ≤ 30.5 mL/kg/min

Exclusion Criteria:

* Estrogen supplementation (in any form) within the previous 6 months
* Any medication that could affect outcome measures such as statins, blood pressure medications, or anti-depressives
* Use of anti-oxidant supplements, in excess of standard multi-vitamins (1 tablet/day) and/or any supplements known to target Nrf2 including resveratrol, Protandim, and sulforaphane
* Current smoker
* Body Mass Index (BMI) greater than 33 kg/m2 (Class I Obesity)
* Any chronic illness that could affect outcome measures, including diabetes, liver or renal disease, or cancer (other than skin cancer)
* History of a myocardial infarction within the last 6 months, clinically significant aortic stenosis, use of cardiac defibrillator, or uncontrolled angina
* Clinically significant arrhythmia on a resting EKG or significant EKG changes during the baseline VO2 max test
* Any other condition that would contraindicate maximal exercise testing, including elevated blood pressure at rest (systolic BP >150 or diastolic BP >90 mm Hg on at least 2 measurements, at least 10 minutes apart) or musculoskeletal problems

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Nrf2 activation in response to acute exercise | Comparing trials separated by one week (supplement vs. placebo)
  Nrf2/ARE Binding Assay

SECONDARY OUTCOMES:
NQO1 gene expression in response to acute exercise | Comparing trials separated by one week (supplement vs. placebo)
  NQO1 mRNA measured with RT-qPCR
HO-1 gene expression in response to acute exercise | Comparing trials separated by one week (supplement vs. placebo)
  HO-1 mRNA measured with RT-qPCR
Glutathione reductase (GR) gene expression in response to acute exercise | Comparing trials separated by one week (supplement vs. placebo)
  GR mRNA measured with RT-qPCR

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Arizona University, Flagstaff, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodriguez DJ, Ostrom EL, Chassman C, Robertson J, Pan V, Buscaglia R, Eggler AL, Traustadottir T. Sulforaphane improves exercise-induced NRF2 signaling in older adults: an in vivo-ex vivo approach. Geroscience. 2025 Oct 16. doi: 10.1007/s11357-025-01939-5. Online ahead of print. PMID 41099966